CLINICAL TRIAL: NCT05980208
Title: A Real-world Study of Inetetamab for First-line Treatment of HER2-positive Inoperable Locally Advanced or Relapsed Metastatic Breast Cancer
Brief Title: A Real-world Study of Inetetamab for First-line Treatment of MBC
Status: Not yet recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Hunan Medical University General Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: KY-2023071101
Record Dates: First submitted 2023-07-24; First posted 2023-08-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Real-world Study
Keywords: breast cancer; real-world study; HER2-postive; inetetamab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inetetamab: Inetetamab-based treatment for first-line treatment of HER2-positive MBC
  Interventions: Drug: Inetetamab

INTERVENTIONS:
Drug: Inetetamab — Inetetamab-based treatment for first-line treatment of HER2-positive MBC

SUMMARY:
This is a prospective, multicenter, real-world study aimed at evaluating the efficacy and safety of inetetamab+chemotherapy or inetetamab+pyrotinib+chemotherapy or inetetamab+pertuzumab+chemotherapy in the treatment of HER2 positive inoperable locally advanced or recurrent metastatic breast cancer. The research results will provide new targeted treatment strategies for HER2 positive breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years and ≤75 years;Patients aged ≥18 years and ≤75 years;
* Her2-positive invasive breast cancer confirmed by pathological examination met the following conditions:

Positive HER2 expression: Immunohistochemical staining (IHC) showed positive HER2 3+ and/or fluorescence in situ hybridization (FISH); Tumor staging: inoperable locally advanced or recurrent metastatic breast cancer; Patients with local recurrence must be confirmed by the investigator to be unable to undergo radical surgical excision.

* At least one measurable lesion was present according to RECIST1.1 criteria;
* The ECOG score is 0 to 1;
* No systematic antitumor therapy (except first-line endocrine therapy) has been received at the locally advanced stage (clinically inoperable) or at the stage of recurrence and metastasis;
* The functional level of major organs must meet the following requirements (no blood transfusion within 2 weeks prior to screening, no use of leukocyte enhancing and platelet enhancing drugs) :

  1. Blood routine: neutrophils (ANC) ≥1.5×109/L; Platelet count (PLT) ≥90×109/L; Hemoglobin (Hb) ≥90 g/L;
  2. Blood biochemistry: total bilirubin (TBIL) ≤ upper limit of normal value (ULN), known patients with Gilbert syndrome, TBIL≤2×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×ULN, patients with liver metastasis required ALT and AST≤5×ULN; Alkaline phosphatase ≤2.5×ULN; Urea/urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN;
  3. Cardiac ultrasound: left ventricular ejection fraction (LVEF) ≥50%;
  4. 12-lead electrocardiogram: Fridericia corrected QT interval (QTcF) <470 msec;
* Expected survival ≥3 months;
* Participate in this study voluntarily, sign informed consent, have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

* Known allergic history of drug components of the program;
* Patients judged unsuitable for systematic chemotherapy by researchers;
* Use of endocrine therapy drugs within 14 days before baseline;
* Patients with only bone or skin as target lesions;
* Other malignancies, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or squamous cell carcinoma, within the previous 5 years;
* Peripheral neuropathy ≥ grade 3 according to CTCAE 5.0 criteria;
* Had received major surgical procedures or significant trauma within 4 weeks prior to randomization, or was expected to receive major surgical treatment;
* Serious heart disease or discomfort, including but not limited to:

heart failure or contraction dysfunction (LVEF <50%) past medical history high risk or the need for treatment of angina or arrhythmia (such as second degree atrioventricular block type 2 or 3 degree atrioventricular block, ventricular tachycardia) clinical significance of heart valve disease ECG showed wall permeability myocardial infarction poorly controlled hypertension, systolic blood pressure>150 mmHg and/or diastolic blood pressure>100 mmHg

* Dysphagia, chronic diarrhea, intestinal obstruction and other factors affecting drug delivery and absorption;
* A history of immunodeficiency, including HIV infection, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;
* Participated in other drug clinical studies within 4 weeks prior to screening;
* There is a third interstitial effusion (such as pleural fluid and ascites) that cannot be controlled by drainage or other methods;
* Pregnant or lactating women, women of childbearing age who are unable to take effective contraceptive measures throughout the trial period;
* Have a serious concomitant disease or other co-medical condition that interferes with planned treatment or any other condition that is not suitable for participation in the study, such as active hepatitis B, lung infection requiring treatment, etc.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: First-line treatment of HER2 positive inoperable local advanced or recurrent metastatic breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The survival time from the date of randomization to the date of the first documented progression or date of death, whichever came first, assessed up to 60 months

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date at the end of the second treatment cycle (42 days)
  The total rate of CR+PR after the completion of two cycles of treatment.
Overall survival | The time from randomization to death from any cause, whichever came first, assessed up to 60 months
  The time from randomization to death from any cause
Adverse Events | The time from randomization to reach the endpoint, assessed up to 60 months
  All adverse events [including adverse events (AE / SAE) and ADR (adverse drug reactions)] will be collected when known. The classification of adverse reactions shall refer to CTCAE5.0 in case of adverse events / reactions. In case of serious adverse events, the investigators must immediately take necessary treatment measures to protect the safety of subjects. All adverse events / reactions should be tracked and observed. If the adverse events have not recovered, the investigator shall continue to give necessary treatment, report and record, and deal with special cases according to the management opinions of relevant departments.

IPD SHARING:
Plan to Share IPD: Undecided